CLINICAL TRIAL: NCT04789304
Title: Safety, Tolerability and Pharmacokinetics of Multiple Rising Oral Doses of BI 1595043 (Double-blind, Randomised, Placebocontrolled, Parallel Group Design) in Healthy Male Subjects
Brief Title: A Study to Test How Healthy Men Tolerate Different Doses of BI 1595043
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1445-0002; 2020-004923-18 (EudraCT Number)
Record Dates: First submitted 2021-03-08; First posted 2021-03-09 (Actual); Results first posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2023-07

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: As this is a Multiple Rising Dose (MRD) trial, blinded individuals will be aware of the current dose level.
  All individuals are unblinded regarding the midazolam administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo / Placebo + Midazolam (Placebo Comparator): Placebo matching BI 1595043. Patients included in the placebo arm corresponding to dose group 3, also received Midazolam.
  Interventions: Drug: Placebo; Drug: Midazolam
- 15 mg BI 1595043 (Experimental): 15 milligram (mg) BI 1595043. Dose group 1.
  Interventions: Drug: BI 1595043
- 30 mg BI 1595043 (Experimental): 30 mg BI 1595043. Dose group 2.
  Interventions: Drug: BI 1595043
- 60 mg BI 1595043 + Midazolam (Experimental): 60 mg BI 1595043 + Midazolam. Dose group 3.
  Interventions: Drug: BI 1595043; Drug: Midazolam

INTERVENTIONS:
Drug: BI 1595043 — BI 1595043
  Arms: 15 mg BI 1595043; 30 mg BI 1595043; 60 mg BI 1595043 + Midazolam
Drug: Placebo — Placebo
  Arms: Placebo / Placebo + Midazolam
Drug: Midazolam — Midazolam
  Arms: 60 mg BI 1595043 + Midazolam; Placebo / Placebo + Midazolam

SUMMARY:
The primary objectives of this trial are to investigate safety and tolerability of BI 1595043 in healthy male subjects following administration of multiple rising doses over 14 days.

Secondary objectives are the exploration of pharmacokinetics (PK) of BI 1595043 after single and multiple dosing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR), body temperature), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 50 years (inclusive)
* BMI of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Male subjects who meet any of the following criteria from at least 30 days before the first administration of trial medication until 30 days after trial completion:

  * Use of adequate contraception, i.e. use of condom (male subjects) plus any of the following methods (female partners): intrauterine device, hormonal contraception (e.g. implants, injectables, combined oral or vaginal contraceptives) that started at least 2 months prior to first drug administration to the male subject, or barrier method (e.g. diaphragm with spermicide), or surgically sterilised (including bilateral tubal occlusion, hysterectomy or bilateral oophorectomy), or postmenopausal, defined as at least 1 year of spontaneous amenorrhea
  * Sexually abstinent
  * Vasectomised (vasectomy at least 1 year prior to enrolment) in combination with a barrier method (i.e. condom) Unprotected sexual intercourse (i.e. without use of condom) with a pregnant female partner and sperm donation is not allowed throughout the study and until 30 days after trial completion

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Further exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A double-blind, randomised, placebo-controlled, parallel group trial to investigate the safety and tolerability of BI 1595043 in healthy male subjects after oral administration of multiple rising doses of 14 days.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they strictly met all inclusion and none of the exclusion criteria. All subjects were informed that they were free to withdraw their consent at any time during the trial without penalty or prejudice. Subjects were recruited to a dose group according to their temporal availability and randomised within each dose group in a 4:1 ratio (trial drug to placebo).
Groups:
- Placebo / Placebo + Midazolam: Film-coated tablets of Placebo, matching to 5 milligram (mg) and 25 mg BI 1595043,were administered orally once daily with 240 milliliter (mL) of water to the corresponding dose group.
  Patients included in the placebo arm corresponding to dose group 3, also received a single oral dose of 75 µg (5 mg/5 mL diluted to 50 µg/mL·1.5 mL) solution for injection of midazolam on Day - 1, Day 1 and Day 18.
- 15 mg BI 1595043 qd: 3 film-coated tablets of 5 milligram (mg) (total dose: 15 mg) BI 1595043 were administered orally once daily (qd), with 240 mL of water after an overnight fast of at least 10 hours (h) on Day 1, followed by a washout of 4 days and from Day 5 to Day 18. Dose group 1.
- 30 mg BI 1595043 qd: 1 film-coated tablet of 5 mg and 1 film-coated tablet of 25 mg (total dose: 30 mg) of BI 1595043 were administered orally once daily (qd), with 240 mL of water after an overnight fast of at least 10 hours (h) on Day 1, followed by a washout of 4 days and from Day 5 to Day 18. Dose group 2.
- 60 mg BI 1595043 qd + Midazolam: 2 film-coated tablets of 5 mg and 2 film-coated tablets of 25 mg (total dose: 60 mg) of BI 1595043 were administered orally once daily (qd), with 240 mL of water after an overnight fast of at least 10 hours (h) on Day 1, followed by a washout of 4 days and from Day 5 to Day 18. On Day - 1, Day 1 and Day 18, 75 µg (5 mg/5 mL diluted to 50 µg/mL·1.5 mL) solution for injection of midazolam was administered as single oral dose. Dose group 3.
Period: Overall Study
Arm/Group | Placebo / Placebo + Midazolam | 15 mg BI 1595043 qd | 30 mg BI 1595043 qd | 60 mg BI 1595043 qd + Midazolam
Started (Treated) | 6 | 8 | 8 | 8
Completed | 6 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): The TS included all subjects who were randomised and treated with at least one dose of trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo / Placebo + Midazolam | 15 mg BI 1595043 qd | 30 mg BI 1595043 qd | 60 mg BI 1595043 qd + Midazolam | Total
Number analyzed (Participants) | 6 | 8 | 8 | 8 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.8 (11.7) | 30.5 (7.8) | 30.6 (7.8) | 40.8 (5.8) | 35.1 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 6 | 8 | 8 | 8 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 8 | 8 | 8 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 8 | 8 | 7 | 29
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Drug-related Adverse Events (AEs)
Description: Percentage of participants with drug-related adverse events (AEs). The causal relationship of AEs to the investigational product was judged by the investigator. The investigator was asked to record a 'yes' if there was, in his/her judgement, a reasonable causal relationship between the investigational product administered and the AE or a 'no' if there was, in his/her judgement, no reasonable causal relationship between the investigational product administered and the AE.
Time Frame: From first drug administration until end of trial examination, up to 30 days.
Population: Treated Set (TS): The TS included all subjects who were randomised and treated with at least one dose of trial drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo / Placebo + Midazolam | 15 mg BI 1595043 qd | 30 mg BI 1595043 qd | 60 mg BI 1595043 qd + Midazolam
Number analyzed (Participants) | 6 | 8 | 8 | 8
Percentage of participants | 0 | 12.5 | 25.0 | 37.5

2. Secondary Outcome: Area Under the Concentration-time Curve of BI 1595043 in Plasma at Steady State Over a Uniform Dosing Interval τ (AUC0-τ,ss)
Description: Area under the concentration-time curve of BI 1595043 in plasma at steady state over a uniform dosing interval τ (AUC0-τ,ss) after the last dose of BI 1595043.
Time Frame: 0.25 hours before and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 34, 48, 72, 96, 120 and 144 hours after the last dose of BI 1595043.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): The PKS included all subjects in the TS who provided at least one PK endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a subject was included in the PKS, even if he/she contributed only one PK parameter value for one period to the statistical assessment. Only participants with non-missing values were included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanomol per Liter
Arm/Group | 15 mg BI 1595043 qd | 30 mg BI 1595043 qd | 60 mg BI 1595043 qd + Midazolam
Number analyzed (Participants) | 8 | 8 | 7
Hours*nanomol per Liter | 1970 (22.1) | 3630 (10.2) | 8170 (18.5)

3. Secondary Outcome: Maximum Measured Concentration of BI 1595043 in Plasma at Steady State Over a Uniform Dosing Interval τ (Cmax,ss)
Description: Maximum measured concentration of BI 1595043 in plasma at steady state over a uniform dosing interval τ (Cmax,ss) after the last dose of BI 1595043.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomol per Liter
Arm/Group | 15 mg BI 1595043 qd | 30 mg BI 1595043 qd | 60 mg BI 1595043 qd + Midazolam
Number analyzed (Participants) | 8 | 8 | 7
Nanomol per Liter | 333 (22.1) | 797 (23.3) | 1630 (36.8)

4. Secondary Outcome: Minimum Measured Concentration of BI 1595043 in Plasma at Steady State Over a Uniform Dosing Interval τ (Cmin,ss)
Description: Minimum measured concentration of BI 1595043 in plasma at steady state over a uniform dosing interval τ (Cmin,ss) after the last dose of BI 1595043.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomole per Liter
Arm/Group | 15 mg BI 1595043 qd | 30 mg BI 1595043 qd | 60 mg BI 1595043 qd + Midazolam
Number analyzed (Participants) | 8 | 8 | 7
Nanomole per Liter | 12.7 (58.6) | 17.7 (13.6) | 36.4 (33.4)

5. Secondary Outcome: Accumulation Ratio Based on Maximum Measured Concentration of BI 1595043 in Plasma at Steady State Over a Uniform Dosing Interval τ (Cmax,ss) (RA, Cmax)
Description: Accumulation ratio based on maximum measured concentration of BI 1595043 in plasma at steady state over a uniform dosing interval τ (Cmax,ss) (RA, Cmax), after the last dose.
  RA,Cmax = Cmax after last dose / Cmax after first dose.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | 15 mg BI 1595043 qd | 30 mg BI 1595043 qd | 60 mg BI 1595043 qd + Midazolam
Number analyzed (Participants) | 8 | 8 | 7
Ratio | 0.894 (19.9) | 1.12 (30.3) | 1.09 (31.4)

6. Secondary Outcome: Accumulation Ratio Based on Area Under the Concentration-time Curve of BI 1595043 in Plasma at Steady State Over a Uniform Dosing Interval τ (AUC0-τ,ss) (RA, AUC)
Description: Accumulation ratio based on area under the concentration-time curve of BI 1595043 in plasma at steady state over a uniform dosing interval τ (AUC0-τ,ss) (RA, AUC).
  RA,AUC = AUC0-\tau after last dose / AUC0-\tau after first dose.
Time Frame: as for outcome 2
Population: Pharmacokinetic (PK) parameter analysis set (PKS): The PKS included all subjects in the TS who provided at least one PK endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a subject was included in the PKS, even if he/she contributed only one PK parameter value for one period to the statistical assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | 15 mg BI 1595043 qd | 30 mg BI 1595043 qd | 60 mg BI 1595043 qd + Midazolam
Number analyzed (Participants) | 8 | 8 | 8
Ratio | 1.04 (4.93) | 1.06 (11.4) | 1.11 (4.97)

ADVERSE EVENTS:
Time Frame: From first drug administration until end of trial examination, up to 30 days.
Description: Treated Set (TS): The TS included all subjects who were randomised and treated with at least one dose of trial drug.
Arm/Group | Placebo / Placebo + Midazolam | 15 mg BI 1595043 qd | 30 mg BI 1595043 qd | 60 mg BI 1595043 qd + Midazolam
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 3/6 | 8/8 | 4/8 | 5/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo / Placebo + Midazolam (N=6) | 15 mg BI 1595043 qd (N=8) | 30 mg BI 1595043 qd (N=8) | 60 mg BI 1595043 qd + Midazolam (N=8)
Eye irritation (Eye disorders) | 0 | 0 | 0 | 2
Blepharitis (Eye disorders) | 0 | 1 | 0 | 0
Lenticular opacities (Eye disorders) | 0 | 1 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 3 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The sponsor decided to terminate the development of BI 1595043 in all indications, the trial prematurely ended according to a protocol-defined option. Trial was completed as described in protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-07-23): https://cdn.clinicaltrials.gov/large-docs/04/NCT04789304/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/04/NCT04789304/SAP_001.pdf